CLINICAL TRIAL: NCT06205563
Title: The Effects of Short-term Supervised High-intensity Interval Training and Moderate Intensity Continuous Training on Weight Loss and Metabolic Indicators in Obese Children Under Energy Limited Balanced Diet
Brief Title: The Therapeutic Effect of Different Exercise Intensities on Weight Loss in Obese Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhu Shunye, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOWL
Record Dates: First submitted 2024-01-03; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss; Obese Children and Adolescents
MeSH Terms: conditions — Weight Loss | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Behavioral: high-intensity interval training
- Arm B (Active Comparator)
  Interventions: Behavioral: moderate intensity continuous training

INTERVENTIONS:
Behavioral: high-intensity interval training — High-intensity interval training (to significantly faster breathing, a significant increase in breathing depth, a significant increase in heart rate, sweating, and the need to stop exercising and adjust your breathing before you can speak; Energy expenditure (METy ≥6.00 in children) : Participants randomly assigned to HIIT will perform a 10-minute warm-up at 60-70% of their maximum heart rate (HRmax). After this, they will walk, run, or bike at 85-95% of their maximum heart rate for four sessions of four minutes each, with three minutes of active recovery (50-70% of their maximum heart rate) in between. The participants were given a five-minute cooling-off period at the end, for a total of 40 minutes of exercise. Participants will be required to participate in supervised exercise classes at least five times and up to seven times a week for 12 weeks. Each participant will be free to wear a smart electronic sports bracelet, which can be used to punch in sports.
  Arms: Arm A
Behavioral: moderate intensity continuous training — Moderate intensity continuous training (rapid breathing, rapid heart rate, slight sweating, but still able to talk easily; Energy expenditure (children METy) 3.00 to 5.99) : Participants randomly assigned to the MICT group will walk, run, or cycle continuously for 40 minutes at 60-70% HRmax. Participants will be required to participate in supervised exercise classes at least five times and up to seven times a week for 12 weeks. Each participant will be free to wear a smart electronic sports bracelet, which can be used to punch in sports.
  Arms: Arm B

SUMMARY:
The incidence of childhood obesity is increasing, followed by metabolic diseases related to overweight and obesity in children. High intensity interval training (HIIT) has recently been shown to improve the body composition and cardiovascular health of obese children. Currently, there is little evidence on the impact of exercise intensity on endocrine and metabolic indicators and quality of life in obese children.

The main purpose of this study is to compare the effects of short-term supervised high-intensity interval training and moderate intensity continuous training (MICT) on metabolic indicators in obese children under an energy limited balanced diet. A multicenter prospective randomized controlled trial was conducted on 388 obese children in South China. The experimental group will be randomly assigned to (1) HIIT and energy limited balanced diet, and (2) MICT and energy limited balanced diet. The experimental group will participate in a 3-month (supervised) exercise training. The measurement of the study endpoint will be followed up at baseline, 3 months (after supervised intervention), 9 months, and 1 year. The primary endpoint is the percentage of weight loss (△ Wt%). Secondary endpoints include waist to height ratio, body mass index (BMI), body fat percentage, insulin resistance index (HOMA-IR), insulin secretion index (ISI), and Δ HtSDSBA. The results of this study will generate a wealth of information on the impact of exercise intensity on weight loss and endocrine metabolism in obese children, and develop more effective evidence-based exercise prescription guidelines in this population.

ELIGIBILITY:
Inclusion Criteria:

1. The guardian understands and signs the informed consent. If the subject is at least 8 years old, the informed consent must be signed.
2. Age 6~16 years old, male and female;
3. BMI≥ "sex-age BMI reference point for obesity screening of school-age children aged 6-18 years";
4. no disability;
5. Joint cardiopulmonary function assessment showed that participation was safe;
6. At least one year of follow-up is expected.

Exclusion Criteria:

1. Have high blood pressure (defined as systolic or diastolic blood pressure values above the 95th percentile), any history or evidence of heart disease and/or abnormal resting or stress echocardiography or a combined cardiopulmonary function assessment indicating that participation is not safe;
2. have any chronic disease, such as chronic asthma, kidney disease, type 1 diabetes, epilepsy, etc.;
3. suffering from organic diseases, such as ovarian tumors, hamartoma, etc.;
4. A smoking habit or orthopedic/neurological condition that may limit exercise ability;
5. Confirmed attention deficit hyperactivity disorder and steroid use.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 388 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
△Wt% | From enrollment to the end of treatment at 12 weeks
  Percentage of weight loss (△Wt%) = (weight at week n - weight at week 0)/weight at week 0 *100%

IPD SHARING:
Plan to Share IPD: Undecided